CLINICAL TRIAL: NCT02385630
Title: Longitudinal Assessment of Gut Hormone Secretion Following Upper Gastrointestinal Surgery for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: University College Dublin (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Surgical Research Fellow, St. James's Hospital, Ireland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CRFSJ 0058; 2014-12 CA (Other: St. James's Hospital Research Ethics Committee)
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Weight Loss; Malnutrition
Keywords: Longitudinal Studies; Esophagectomy; Gastrectomy; Hunger; Appetite; Glucagon-like Peptide 1; Peptide YY; Ghrelin; Satiety Response; Feeding Behavior; Meals; Postprandial Period
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Weight Loss; Malnutrition; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esophagectomy (Experimental): Serial assessment:
  Fasting gut hormones, post-prandial gut hormone response to a standardized 400kcal meal
  Interventions: Other: Standardized 400kcal semi-liquid meal
- Gastrectomy (Experimental): Serial assessment:
  Fasting gut hormones, post-prandial gut hormone response to a standardized 400kcal meal
  Interventions: Other: Standardized 400kcal semi-liquid meal

INTERVENTIONS:
Other: Standardized 400kcal semi-liquid meal — Used to assess post-prandial gut hormone response pre-operatively and at 10 days, 4 weeks, 6 months and 12 months post-operatively.

SUMMARY:
Surgery is the cornerstone of treatment for patients with oesophageal or gastric cancer, but while surgical removal of the tumour (oesophagectomy or gastrectomy) may offer the best chance of cure, these are major operations associated with specific long term complications. Weight loss and poor nutrition are relatively common problems among patients who attain long-term cancer remission and cure after surgery. The mechanisms underlying these problems are not well understood and therefore treatment options are limited.

The investigators research has demonstrated increased levels of chemical messengers (gut hormones) released from the gastrointestinal tract after meals in patients who have previously undergone upper gastrointestinal surgery. These chemical messengers play a role in signalling the feeling of fullness during and after a meal (satiety). Understanding the mechanisms involved in increased gut hormone secretion after these operations may allow us to use certain medications to block gut hormone release and hence reduce satiety allowing patients to eat more, regain weight and prevent nutritional complications after surgery.

Exaggerated post-prandial satiety gut hormone responses following oesophagectomy have, however, only been established cross-sectionally and therefore the time course for development of increased gut hormone secretion is unknown. Data collected from this study will provide important information about optimal timing of therapeutic intervention in this patient group, while offering mechanistic insights with regard to the pathophysiologic process underlying post-operative early satiety.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo two-stage, three-stage or transhiatal oesophagectomy with gastric conduit reconstruction OR total gastrectomy with Roux-en-Y reconstruction

Exclusion Criteria:

1. Significant and persistent chemoradiotherapy complication
2. Other previous upper gastrointestinal surgery
3. Unwell or unable to eat
4. Other disease or medications which may affect satiety gut hormone responses
5. Active and significant psychiatric illness including substance misuse
6. Cognitive or communication issues or any factors affecting capacity to consent to participation
7. History of significant food allergy, certain dietary restrictions
8. Confirmed or suspected residual or recurrent disease after surgery, synchronous or metachronous malignancy
9. Significant surgical complication, aspiration risk or deterioration in performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Post-prandial satiety gut hormone area under the curve | 1 year

SECONDARY OUTCOMES:
Body anthropometry | 1 year
  Weight (kg)
EORTC health related quality of life at one year | 1 year
  Global health status score
Subjective symptom scores | 1 year
  Sigstad dumping score
Fasting ghrelin concentration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MCh, FRCS, Principal Investigator — Department of Surgery, St. James's Hospital
Locations (1):
- Wellcome Trust-Health Research Board Clinical Research Facility, St. James's Hospital, Dublin, Ireland

REFERENCES:
- [Background] Martin L, Lagergren J, Lindblad M, Rouvelas I, Lagergren P. Malnutrition after oesophageal cancer surgery in Sweden. Br J Surg. 2007 Dec;94(12):1496-500. doi: 10.1002/bjs.5881. PMID 17668914
- [Background] Martin L, Lagergren P. Long-term weight change after oesophageal cancer surgery. Br J Surg. 2009 Nov;96(11):1308-14. doi: 10.1002/bjs.6723. PMID 19847871
- [Background] Donohoe CL, McGillycuddy E, Reynolds JV. Long-term health-related quality of life for disease-free esophageal cancer patients. World J Surg. 2011 Aug;35(8):1853-60. doi: 10.1007/s00268-011-1123-6. PMID 21553202
- [Background] Yamamoto K, Takiguchi S, Miyata H, Adachi S, Hiura Y, Yamasaki M, Nakajima K, Fujiwara Y, Mori M, Kangawa K, Doki Y. Randomized phase II study of clinical effects of ghrelin after esophagectomy with gastric tube reconstruction. Surgery. 2010 Jul;148(1):31-8. doi: 10.1016/j.surg.2009.11.026. Epub 2010 Jan 21. PMID 20096432
- [Background] Miyazaki T, Tanaka N, Hirai H, Yokobori T, Sano A, Sakai M, Inose T, Sohda M, Nakajima M, Fukuchi M, Kato H, Kuwano H. Ghrelin level and body weight loss after esophagectomy for esophageal cancer. J Surg Res. 2012 Jul;176(1):74-8. doi: 10.1016/j.jss.2011.09.016. Epub 2011 Oct 3. PMID 22137988
- [Background] Koizumi M, Hosoya Y, Dezaki K, Yada T, Hosoda H, Kangawa K, Nagai H, Lefor AT, Sata N, Yasuda Y. Postoperative weight loss does not resolve after esophagectomy despite normal serum ghrelin levels. Ann Thorac Surg. 2011 Apr;91(4):1032-7. doi: 10.1016/j.athoracsur.2010.11.072. PMID 21440118
- [Background] Doki Y, Takachi K, Ishikawa O, Miyashiro I, Sasaki Y, Ohigashi H, Nakajima H, Hosoda H, Kangawa K, Sasakuma F, Motoori M, Imaoka S. Ghrelin reduction after esophageal substitution and its correlation to postoperative body weight loss in esophageal cancer patients. Surgery. 2006 Jun;139(6):797-805. doi: 10.1016/j.surg.2005.11.015. PMID 16782437
- [Background] le Roux CW, Welbourn R, Werling M, Osborne A, Kokkinos A, Laurenius A, Lonroth H, Fandriks L, Ghatei MA, Bloom SR, Olbers T. Gut hormones as mediators of appetite and weight loss after Roux-en-Y gastric bypass. Ann Surg. 2007 Nov;246(5):780-5. doi: 10.1097/SLA.0b013e3180caa3e3. PMID 17968169
- [Background] Papamargaritis D, le Roux CW, Sioka E, Koukoulis G, Tzovaras G, Zacharoulis D. Changes in gut hormone profile and glucose homeostasis after laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2013 Mar-Apr;9(2):192-201. doi: 10.1016/j.soard.2012.08.007. Epub 2012 Aug 24. PMID 23183113
- [Background] Miholic J, Orskov C, Holst JJ, Kotzerke J, Pichlmayr R. Postprandial release of glucagon-like peptide-1, pancreatic glucagon, and insulin after esophageal resection. Digestion. 1993;54(2):73-8. doi: 10.1159/000201016. PMID 8319842
- [Background] le Roux CW, Borg C, Wallis K, Vincent RP, Bueter M, Goodlad R, Ghatei MA, Patel A, Bloom SR, Aylwin SJ. Gut hypertrophy after gastric bypass is associated with increased glucagon-like peptide 2 and intestinal crypt cell proliferation. Ann Surg. 2010 Jul;252(1):50-6. doi: 10.1097/SLA.0b013e3181d3d21f. PMID 20562614
- [Result] Elliott JA, Docherty NG, Eckhardt HG, Doyle SL, Guinan EM, Ravi N, Reynolds JV, Roux CWL. Weight Loss, Satiety, and the Postprandial Gut Hormone Response After Esophagectomy: A Prospective Study. Ann Surg. 2017 Jul;266(1):82-90. doi: 10.1097/SLA.0000000000001918. PMID 27455150
- [Result] Elliott JA, Docherty NG, Murphy CF, Eckhardt HG, Doyle SL, Guinan EM, Ravi N, Reynolds JV, le Roux CW. Changes in gut hormones, glycaemic response and symptoms after oesophagectomy. Br J Surg. 2019 May;106(6):735-746. doi: 10.1002/bjs.11118. Epub 2019 Mar 18. PMID 30883706
- See also: Wellcome Trust-HRB Clinical Research Facility — http://www.sjhcrf.ie